CLINICAL TRIAL: NCT00643409
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Levofloxacin for the Treatment of Acute Bacterial Maxillary Sinusitis in Adults Undergoing Diagnostic Sinus Aspiration
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Trial of Azithromycin SR Compared With Levofloxacin for the Treatment of Sinus Infections in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661078
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis | interventions — Azithromycin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: azithromycin SR (Zithromax; compound: CP-62,993); Other: placebo
- 2 (Experimental)
  Interventions: Drug: levofloxacin; Other: placebo

INTERVENTIONS:
Drug: azithromycin SR (Zithromax; compound: CP-62,993) — Azithromycin SR 2.0 g by mouth in the form of a slurry x 1 dose
  Arms: 1
Other: placebo — placebo
  Arms: 1
Drug: levofloxacin — levofloxacin 500 mg capsule by mouth qd x 10 days
  Arms: 2
Other: placebo — placebo
  Arms: 2

SUMMARY:
The objectives of the study were to confirm that a single, 2.0-g dose of azithromycin sustained release (SR) was at least as effective to 10 days of oral levofloxacin 500 mg once a day, when used to treat adults with uncomplicated, acute bacterial sinus infections, and to evaluate the safety of both treatments.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they had a clinical diagnosis of acute bacterial maxillary sinusitis as demonstrated by presence of the cardinal signs and symptoms for a minimum duration of 7 days, a sinus X-ray (Water's view) confirming the clinical diagnosis of maxillary sinusitis, and 2 or more of following: fever, leukocytosis, frequent coughing, headache, nasal congestion, or post-nasal drainage.

Exclusion Criteria:

Patients were excluded if they were treated with any systemic antibiotic within 7 days prior to enrollment, had symptoms lasting for longer than 28 days, had 4 or more episodes of acute sinusitis within the preceding 12 months, had nasal or sinus surgery within 3 months prior (except for a diagnostic procedure), or complicated or nosocomial sinusitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2003-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
sponsor assessment of clinical response for the Clinical per Protocol population | Test of Cure (TOC) visit (Day 17-24)

SECONDARY OUTCOMES:
sponsor assessment of clinical response by baseline pathogen for the Bacteriological per Protocol population | EOT visit and TOC visit
investigator assessment of clinical response for the Clinical per Protocol population | TOC visit
bacteriological response on a per pathogen basis for the Bacteriological Per Protocol population | TOC visit
summary of baseline susceptibilities | Study endpoint
adverse events | Continuous
laboratory abnormalities | during and post-treatment
sponsor assessment of clinical response for the Clinical per Protocol population | End of Treatment (EOT) visit (Day 11-13)
sponsor assessment of clinical response for the remaining study populations | EOT visit and TOC visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- United States (40):
  - Pfizer Investigational Site, Alabaster, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Hueytown, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Pelham, Alabama
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Clovis, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Bridgeport, Connecticut
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, Richland, Michigan
  - Pfizer Investigational Site, Three Rivers, Michigan
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Missoula, Montana
  - Pfizer Investigational Site, Charlote, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Morrisville, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Plymouth Meeting, Pennsylvania
  - Pfizer Investigational Site, Orangeburg, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Amarillo, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Pasadena, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
- Pfizer Investigational Site, Buenos Aires, Argentina
- Pfizer Investigational Site, Santiago, Chile
- Costa Rica (5):
  - Pfizer Investigational Site, Bo. Aranjuez, Provincia de San José
  - Pfizer Investigational Site, Escazú, Provincia de San José
  - Pfizer Investigational Site, Guadalupe, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
  - Pfizer Investigational Site, Uruca, Provincia de San José
- Pfizer Investigational Site, Prague, Czechia
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- Pfizer Investigational Site, Rostock, Germany
- India (3):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Pfizer Investigational Site, Vilnius, Lithuania
- Pfizer Investigational Site, Chihuahua City, Chihuahua, Mexico
- Poland (4):
  - Pfizer Investigational Site, Bielsko-Biala
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Poznan
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Košice, Slovakia
  - Pfizer Investigational Site, Martin, Slovakia
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661078&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Trial%20of%20Azithromycin%20SR%20Compared%20with%20Levofloxacin%20for%20the%20Treatment%20of%20Sinus%20I